CLINICAL TRIAL: NCT03179319
Title: Mobile-Based Application "MyChoices" to Increase Uptake of HIV Testing, Detection of New HIV Infections, and Linkage to Care and Prevention Services by Young Men Who Have Sex With Men
Brief Title: Mobile-Based Application "MyChoices"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: University of North Carolina (Other); Montefiore Medical Center (Other); Emory University (Other); Brown University (Other)
Responsible Party: Principal Investigator, Kenneth H. Mayer, MD, Principal Investigator, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U19HD089881 (SubProject 8784); 1U19HD089881 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: HIV; Sexually Transmitted Diseases; Pre-exposure Prophylaxis; Risk Reduction
Keywords: PrEP; HIV testing; Sexually transmitted disease (STD) testing; Mobile app; Young men who have sex with men; Technology
MeSH Terms: conditions — Sexually Transmitted Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyChoices (Experimental): Access to the MyChoices mobile app which includes the HIV test plan with reminders, STI information, PrEP resources, links to testing and PrEP sites, and geo-location features.
  Interventions: Behavioral: MyChoices
- Standard of Care (No Intervention): Participants in this study arm will receive local standard of care for linkage to PrEP and HIV/STI testing.

INTERVENTIONS:
Behavioral: MyChoices — Access to the MyChoices mobile app which includes the HIV test plan with reminders, STI information, PrEP resources, links to testing and PrEP sites, and geo-location features.
  Arms: MyChoices

SUMMARY:
This study is testing the acceptability and feasibility of MyChoices, a mobile application (app), to promote HIV testing and pre-exposure prophylaxis (PrEP) uptake among young men who have sex with men (YMSM).

DETAILED DESCRIPTION:
"MyChoices", an app adapted from HealthMindr and developed using iterative feedback from youth, is being refined to to maximize acceptability among YMSM. "MyChoices" was guided by the Social Cognitive Theory (SCT) model and includes three major functions that are designed to promote self-efficacy, self-regulation, goal-setting and environmental influences in order to impact behavior change. (1) Tracking and Self-Monitoring HIV Risk: In order to target self-regulation, brief surveys within the app are used to assess behavioral patterns of YMSM, particularly around sexual relationships, which are then used to help customize the app for each user. (2) HIV and sexually transmitted infection (STI) Prevention Information: In order to improve self-efficacy for HIV testing and HIV prevention overall, quizzes and infographics that appeal to YMSM have been incorporated into the app, focusing on promotion of HIV prevention and regular HIV testing. The app also allows users to order OraQuick HIV home testing kits and STI home collection kits (for rectal and urethral gonorrhea and Chlamydia and syphilis). Additionally, the app includes information on testing sites and local PrEP clinics (e.g., telephone, address, hours of testing, etc), and external links to specific site webpages that are near the user (determined using GPS technology). (3) HIV Testing Plan: Acknowledging the central role of goal setting and environmental influences on health behavior, the app allows users to create a HIV testing plan by allowing them to compare and choose different screening options (e.g., home self-testing, antigen, rapid). Questions about HIV transmission behaviors and testing history are then asked to create a tailored testing plan. After a HIV testing plan is developed, users have the option to customize reminders for the timeframe selected (e.g., user is pinged every 3 months as a reminder to get tested). Users are able to select from a list of phrases or create their own to ensure privacy. Moreover, geofencing technology allows users to be notified when in the vicinity of testing locations, based on the Geo Positioning System (GPS) location, during the testing timeframe.

This study is part of the iTech NIH U19, which has an overall goal to develop innovative technology-focused interventions addressing the HIV prevention and care continuum for youth.

ELIGIBILITY:
Inclusion Criteria:

* No HIV test in the past 3 months (self-reported).
* Not known to be HIV-infected (self-reported).
* Not currently taking PrEP (self-report).
* Owns or leases a phone with Android platform (for Aims 2 and 3) or iOS platform (Aim 3 only), has an active data plan, and willing to download the MyChoices application.
* Willing to attend an in-person baseline study visit in Boston or the Bronx and complete online follow-up visits.
* Able to understand, read, and speak English.
* Participants ages 15-18: self-report at least one episode of anal intercourse with a male or transfemale partner during the last 6 months.
* Participants ages 19-24: self-report evidence of high risk for acquiring HIV infection including at least one of the following:

  1. at least one episode of condomless anal intercourse with an HIV-infected or unknown HIV status male or transfemale partner during the last 6 months; or
  2. anal intercourse with 2 or more male or transfemale sex partners during the last 6 months; or
  3. exchange of money, gifts, shelter, or drugs for anal sex with a male or transfemale partner during the last 6 months; or
  4. sex with a male or transfemale partner and has had an STI during the last 6 months.

Exclusion Criteria:

* Any health condition that may interfere with participation or the ability to provide informed consent, including any debilitating or life-threatening conditions.
* Prior enrollment in an HIV vaccine trial with receipt of experimental vaccine product and evidence of vaccine-induced seropositivity.
* Known to be HIV-infected.
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender male
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie B Biello, PhD, MPH, Principal Investigator — Protocol Co-Chair, Research Study MPI; Kenneth H Mayer, MD, Principal Investigator — Fenway Health Center
Locations (2):
- United States (2):
  - Fenway Health Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available to outside individuals through contacting the multiple principal investigators (MPIs) at two different times. The first will be after all of the baseline data is collected. The investigators will institute a concept plan process where internal study staff first have the availability to write primary papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, the investigators will welcome this collaboration. A similar process will happen for outcome data; however this will not be possible until the publication and release of the outcome paper(s). Information regarding the availability of data for analysis will be listed on the MPIs' web pages. Contact information for the MPIs will be listed in all manuscripts and publications as another means to access data.

REFERENCES:
- [Derived] Biello KB, Hill-Rorie J, Valente PK, Futterman D, Sullivan PS, Hightow-Weidman L, Muessig K, Dormitzer J, Mimiaga MJ, Mayer KH. Development and Evaluation of a Mobile App Designed to Increase HIV Testing and Pre-exposure Prophylaxis Use Among Young Men Who Have Sex With Men in the United States: Open Pilot Trial. J Med Internet Res. 2021 Mar 24;23(3):e25107. doi: 10.2196/25107. PMID 33759792

RESULTS

PARTICIPANT FLOW:
Groups:
- MyChoices: Access to the MyChoices mobile app which includes the HIV test plan with reminders, STI information, PrEP resources, links to testing and PrEP sites, and geo-location features.
  Participants in this study arm will also receive local standard of care for linkage to PrEP and HIV/STI testing.
Period: Overall Study
Arm/Group | MyChoices | Standard of Care
Started | 40 | 20
3 Month Visit | 37 | 20
Completed (6-month follow up) | 34 | 20
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MyChoices | Standard of Care | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.25 (2.08) | 21.95 (2.26) | 21.48 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 20 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 34 | 17 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 29 | 9 | 38
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Boston, MA | 20 | 10 | 30
  United States: Bronx, NY | 6 | 4 | 10
  United States: Chapel Hill, NC | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Acceptability: System Usability Scale
Description: System Usability Scale: a validated scale that assesses subjective usability of a system, or, in this case, an app. The System Usability Scale consists of a 10 item questionnaire with five response options; from Strongly agree to Strongly disagree. The items scores are converted into a score from 0 (negative) to 100 (positive). A score of ≥50 indicates that the app is acceptable, and a score above 68 is considered above average.
Time Frame: 3 months
Population: Given that this measure is directly related to the MyChoices app, only those who were randomized to the MyChoices app arm were eligible to respond to this outcome; One person had missing data for this item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyChoices
Number analyzed (Participants) | 36
score on a scale | 75.76 (10.72)

2. Primary Outcome: Feasibility: Frequency of Logins
Description: Number of individuals who logged into app at least one time after set up
Time Frame: 3 months
Population: Error in paradata collection resulted in missing app data for 7 participants
Measure: Count of Participants; unit: Participants
Arm/Group | MyChoices
Number analyzed (Participants) | 33
Participants | 31

3. Secondary Outcome: Preliminary Efficacy: Number of Participants Self-reported Having Tested for HIV
Description: Self-report having tested for HIV over follow up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MyChoices | Standard of Care
Number analyzed (Participants) | 38 | 20
Participants | 27 | 13

4. Secondary Outcome: Preliminary Efficacy: Number of Participants Self-reported Having Initiated PrEP
Description: Self-report of participants reporting PrEP initiation anytime over study follow up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MyChoices | Standard of Care
Number analyzed (Participants) | 38 | 20
Participants | 3 | 3

5. Secondary Outcome: Number of Times Participants Used Distinct App Components
Description: The total number of times that participants selected distinct components (e.g., testing plan, ordering, FAQs) of the app were summed
Time Frame: 3 months
Population: Given that this measure is directly related to the MyChoices app, only those who were randomized to the MyChoices app arm were eligible to respond to this outcome. Due to data collection error in the app (which was subsequently fixed), we are missing data from 7 participants.
Measure: Mean (Standard Deviation); unit: App components used
Arm/Group | MyChoices
Number analyzed (Participants) | 33
App components used | 100.58 (86.09)

6. Secondary Outcome: App Content and Functionality Most Utilized
Description: We a priori identified the primary app components (i.e., HIV test plan, location search, ordering supplies, FAQs) and report the number of participants using these app components at least once over follow up
Time Frame: 3 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | MyChoices
Number analyzed (Participants) | 33
Participants
  HIV test plan | 30
  Location search | 26
  FAQs | 22
  Ordering supplies | 31

7. Secondary Outcome: Number of HIV Home Testing Kits Ordered
Description: Number of Participants who ordered at least one HIV home testing kit over follow up
Time Frame: 6 months
Population: Given that this measure is directly related to the MyChoices app, only those who were randomized to the MyChoices app arm were eligible to respond to this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | MyChoices
Number analyzed (Participants) | 40
Participants | 25

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected for 6 months. Across the study, AE data was collected from 11/13/2018 through 11/05/2019.
Arm/Group | MyChoices | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03179319/Prot_SAP_000.pdf